CLINICAL TRIAL: NCT00420147
Title: Effect of In-shoe Wedges on Knee Osteoarthritis
Brief Title: Wedged Orthoses and Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Todd D. Royer, Associate Professor, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P20RR16458-3; P20RR016458 (NIH)
Record Dates: First submitted 2007-01-05; First posted 2007-01-09 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-04

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; orthosis; wedge; gait
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wedged Orthosis (Experimental): Subjects were given a wedged inshoe orthosis
  Interventions: Device: wedged inshoe orthosis
- Neutral Orthosis (Placebo Comparator): Subjects were given a neutral inshoe orthosis.
  Interventions: Device: neutral inshoe orthosis

INTERVENTIONS:
Device: wedged inshoe orthosis — Treatment subjects were prescribed an inshoe wedged orthosis
  Arms: Wedged Orthosis
Device: neutral inshoe orthosis — Control subjects were prescribed a neutral inshoe orthosis
  Arms: Neutral Orthosis

SUMMARY:
The five-year goal of this project is to investigate the effect of in-shoe wedged orthoses on lower extremity function in patients with knee osteoarthritis. In general, our aims address the long-term effects of orthoses. The investigators hypothesize that subjects who use the lateral wedged in shoe orthosis will result in altered gait mechanics that reflect a reduction in the frontal plane knee joint moment compared to subjects who use a neutral in shoe orthosis.

DETAILED DESCRIPTION:
Introduction: In shoe wedged orthoses have been shown to be an effective conservative approach in reducing pain in patients with osteoarthritis (OA). The mechanism responsible for this pain reduction is not well-understood. It is not known whether placing a medial or lateral wedge in the shoe results in alterations in lower extremity alignment, knee joint moments or some combination of the two. The longterm effects of this intervention on OA patients' functional status as well the progression of their OA has not been studied. Therefore, the purpose of this study is to examine the effect of in-shoe wedged orthoses in patients with knee OA on the frontal plane knee joint moment. Methods: 38 patients between the ages of 40-70 yrs with knee OA (grades I-IV) will be recruited from within the medical community. Subjects with a diagnosis of unilateral knee OA of greater than 3 months duration, as defined by the American College of Rheumatology Guidelines, will be included. 19 subjects will be assigned to a treatment group and 19 subjects will be assigned to a control group. The treatment group will receive custom molded orthotics with a lateral wedge. Both the treatment and control groups will be tested initially and then again 1 year later. The dependent variable is peak knee adduction moment. Statistics: A two-way ANOVA will be used to test the hypothesis. This design will include 2 levels of group (control and treatment) and two levels of trial (pretest and 1 yr posttest). Significance will be determined at a level of p<.05.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed unilateral knee osteoarthritis by a qualified physician
* Recent (within 3 months of entrance into the study) radiographic confirmation of OA grade (I-IV) as evidenced by joint space narrowing and the presence of osteophytes
* A score of 50-90 mm on a 100 mm visual analogue pain scale for walking
* Ability to walk independently without the use of assistive devices

Exclusion Criteria:

* History of lower extremity joint surgery or other lower extremity injury that would hinder ambulation
* Severe foot deformity that would prevent the accommodation of the wedged orthotic device
* Other disease process such as neurologic, cardiac, or oncologic, that would hinder one's ability to ambulate
* Any condition, such as diabetes, that results in loss of sensation in the lower extremities

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2002-02; Primary Completion 2006-02 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Royer, PhD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Medial Knee OA - Control: These subjects have tibio-femoral medial knee compartment osteoarthritis and were prescribed a neutral in shoe orthosis
- Medial Knee OA - Treatment: These subjects have tibio-femoral medial knee compartment osteoarthritis and were prescribed a laterally wedged in shoe orthosis
Period: Overall Study
Arm/Group | Medial Knee OA - Control | Medial Knee OA - Treatment
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Medial Knee OA - Control: These subjects have tibio-femoral medial knee compartment osteoarthritis and wore a neutral (non-wedged) in-shoe orthosis as their treatment.
- Medial Knee OA - Treatment: These subjects have tibio-femoral medial knee compartment osteoarthritis and wore a wedged in-shoe orthosis as their treatment.
- Total: Total of all reporting groups
Arm/Group | Medial Knee OA - Control | Medial Knee OA - Treatment | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 12 | 22
  >=65 years | 9 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (9.6) | 62.0 (7.4) | 62.4 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 8 | 9 | 17
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Knee Adduction Moment at Baseline
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Nm/(kg-m)
Groups:
- Medial Knee OA - Control; Medial Knee OA - Treatment: These subjects have tibio-femoral medial knee compartment osteoarthritis
Arm/Group | Medial Knee OA - Control | Medial Knee OA - Treatment
Number analyzed (Participants) | 19 | 19
Nm/(kg-m) | 0.376 (0.118) | 0.342 (0.131)

2. Primary Outcome: Knee Adduction Moment After 12 Months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Nm/(kg-m)
Arm/Group | Medial Knee OA - Control | Medial Knee OA - Treatment
Number analyzed (Participants) | 19 | 19
Nm/(kg-m) | 0.408 (0.108) | 0.358 (0.127)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Medial Knee OA - Control: These subjects have tibio-femoral medial knee compartment osteoarthritis. They were prescribed and wore a neutral in-shoe orthosis.
- Medial Knee OA - Treatment: These subjects have tibio-femoral medial knee compartment osteoarthritis. They were prescribed and wore a laterally wedged in-shoe orthosis.
Arm/Group | Medial Knee OA - Control | Medial Knee OA - Treatment
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

LIMITATIONS AND CAVEATS:
Compliance with the wedged orthoses was self reported by the subjects. There was difficulty with the larger degrees of wedging (10-15 degrees) fitting into the footwear.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No